CLINICAL TRIAL: NCT07403292
Title: Comparative Effects of McGill and McKenzie Exercises on Pain, Range of Motion and Disability in Patients With Chronic Mechanical Low Back Pain
Brief Title: Comparative Effects of McGill and McKenzie Exercises in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0179
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Mechanical Low Back Pain
Keywords: McGill exercises; McKenzie Exercises; pain; range of motion; disability; chronic mechanical low back pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McGill Exercises (Experimental)
  Interventions: Other: McGill Exercises; Other: Standardized Physiotherapy Treatment
- McKenzie Exercises (Active Comparator)
  Interventions: Other: McKenzie Exercises; Other: Standardized Physiotherapy Treatment

INTERVENTIONS:
Other: McGill Exercises — McGill Big three exercises for 10 repetitions and 5-10 seconds of hold initially. Progression was tailored as per the patient's requirements and stamina.
  * Standardized physiotherapy treatment at the first session.
  * McGill curl-up
  * Isometric horizontal side support, either with support on knees or on foot, according to patient stamina.
  * Single leg extension holds on hands and knees, also known as McGill Birddog, either with or without raising the contralateral arm as per patient stamina.
  Arms: McGill Exercises
Other: McKenzie Exercises — McKenzie extension exercise plan (EEP) for 10 repetitions and 5-10 seconds of hold initially. Progression was tailored as per the patient's requirements and symptoms
  * Standardized physiotherapy treatment at the first session.
  * Lying face down in extension on elbows.
  * Full press up.
  * Extension in standing.
  Arms: McKenzie Exercises
Other: Standardized Physiotherapy Treatment — * Electrical Heating Pad was applied for 10 minutes.
  * TENS was applied (low frequency) for 10 minutes.
  * Posterior to Anterior Glides of Lumbar Spine in Maitland Grade-III, with 4 sets and 4 repetitions each. The patient will be in a prone position.

SUMMARY:
The study was conducted to determine the comparative effects of McGill and McKenzie exercises on pain, range of motion and disability in patients with chronic mechanical low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Patients between 20-40 years.
* At least 6 months of history of chronic mechanical low back pain.
* Negative Lasegue's Test.
* Negative Slump Test.
* Patient presenting with NPRS values of above 1 and equal to or less than 6.
* ODI score from 5-24, with the patient showing minimal to moderate disability.
* Patient showing restricted lumbar range of motion in any direction of flexion, extension, and lateral flexion.
* Participants must demonstrate an extension directional preference during clinical examination (For the safety purpose of the patients)

Exclusion Criteria:

* Lumbar radiculopathy.

  * Previous record showing Trauma or accident.
  * Any previous surgical record of Lumbar Spine Surgery.
  * Acute or Subacute low back pain.
  * History of spinal osteoporosis.
  * Vertebral Fractures.
  * Tumors and active infections.
  * Diagnosed psychological disorders.
  * Any spinal deformity
  * Participants who do not show directional preference towards extension

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to the end of the treatment at 6 weeks
  Pain intensity was measured using the Numeric Pain Rating Scale which is abbreviated as NPRS. In this tool, individuals score their pain levels on a scale from 0 to 10. When a participant selects 0, it means they had no pain. On the other hand, if it is 10, the participant must be going through the worst pain imaginable.
Oswestry Disability Index | From enrollment to the end of the treatment at 6 weeks.
  The Oswestry Disability Index (ODI) is a questionnaire that participants fill themselves based on self-reporting. It is based on disability caused by low back pain. Pynsent in Oswestry, England, introduced it in 1980. It has become one of the most widely used and trusted tools for evaluating disability related to back pain.
Lumbar Range of Motion | From enrollment to the end of the 6 weeks
  Different instruments are used in physiotherapy to measure the range of motions, like a goniometer and an inclinometer. An inclinometer is used to measure spinal ROM.

SECONDARY OUTCOMES:
Lumbar Flexion | From enrollment to end of the treatment at 6 weeks.
  Measured by inclinometer.
Lumbar Extension | From enrollment to end of the treatment by 6 weeks.
  Measured by Inclinometer
Lumbar Right Lateral Flexion | From enrollment to the end of 6 weeks
  Measured by Inclinometer
Lumbar Left Lateral Flexion | From enrollment to end of the treatment by 6 weeks.
  Measured by using Inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Shakil ur Rehman, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- Naseer Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabourin S, Tram J, Sheldon BL, Pilitsis JG. Defining minimal clinically important differences in pain and disability outcomes of patients with chronic pain treated with spinal cord stimulation. Journal of Neurosurgery: Spine. 2021;35(2):243-50.
- [Background] Young I, Dunning J, Escaloni J, Maselli F, Prall J, Mourad F, et al. Reliability, construct validity, responsiveness and minimum clinically important difference of the numeric pain rating scale and shoulder pain and disability index in patients with subacromial pain syndrome. Musculoskeletal Science and Practice. 2025:103372.
- [Background] na Fisioterapia MM. Methods & protocols.
- [Background] McGill SM. Low Back Exercises: Evidence for Improving Exercise Regimens. Physical Therapy. 1998;78(7):754-65.
- [Background] Saur PM, Ensink F-BM, Frese K, Seeger D, Hildebrandt J. Lumbar range of motion: reliability and validity of the inclinometer technique in the clinical measurement of trunk flexibility. Spine. 1996;21(11):1332-8.
- [Background] Grotle M, Brox JI, Vøllestad NK. Cross-cultural adaptation of the Norwegian versions of the Roland-Morris Disability Questionnaire and the Oswestry Disability Index. Journal of rehabilitation medicine. 2003;35(5):241-7.
- [Background] JD C. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine. 2005;30:686-96.
- [Background] Alhakami AM, Davis S, Qasheesh M, Shaphe A, Chahal A. Effects of McKenzie and stabilization exercises in reducing pain intensity and functional disability in individuals with nonspecific chronic low back pain: a systematic review. Journal of physical therapy science. 2019;31(7):590-7.
- [Background] Nayyab I, Ghous M, Shakil Ur Rehman S, Yaqoob I. The effects of an exercise programme for core muscle strengthening in patients with low back pain after Caesarian-section: A single blind randomized controlled trial. J Pak Med Assoc. 2021;71(5):1319-25.
- [Background] Ahmed R, Shakil-ur-Rehman S, Sibtain F. Comparison between specific lumber mobilization and core-stability exercises with core-stability exercises alone in mechanical low back pain. Pakistan journal of medical sciences. 2014;30(1):157.
- [Background] Golzar J, Noor S, Tajik O. Convenience sampling. International Journal of Education & Language Studies. 2022;1(2):72-7.
- [Background] Javaherian M, Bashardoust TS, ATTARBASHI MB, KESHTKAR A, Azizi M. Immediate effects of Maitland mobilization and Mulligan techniques on flexion and extension range of motion in patients with chronic nonspecific low back pain: a randomized pilot study. 2017.
- [Background] Waqqar S, Shakil-Ur-Rehman S, Ahmad S. McKenzie treatment versus mulligan sustained natural apophyseal glides for chronic mechanical low back pain. Pak J Med Sci. 2016 Mar-Apr;32(2):476-9. doi: 10.12669/pjms.322.9127. PMID 27182265
- [Background] Kleine-Borgmann J, Schmidt K, Hellmann A, Bingel U. Effects of open-label placebo on pain, functional disability, and spine mobility in patients with chronic back pain: a randomized controlled trial. Pain. 2019;160(12):2891-7.
- [Background] Ghasemi G, Goharjoo M, Faizi M. Effects of conventional core stability and core stability suspension exercises on multifidus muscle endurance, pain and quality of life in people with nonspecific chronic low back pain. Jundishapur Scientific Medical Journal. 2020;18(6):571-84.
- [Background] Hernándeza DMG, Pérez SMO, Ardón FB, Núñez CLT, Moreno JGO. Effectiveness of neurodynamic mobilization and MCGILL-type strengthening exercises in patients with piriformis syndrome: study protocol for a randomized controlled trial. Physical Rehabilitation and Recreational Health Technologies. 2024;9(3):188-200.
- [Background] Purushothaman S, Gayathri K, Thiyagarajan A, Vardhini CI, Babu LH, Nainar M. Clinical Evaluation of the McGill Stabilization Exercise Program for Chronic Nonspecific Low Back Pain: Insights from Case Studies. Journal of Society of Indian Physiotherapists. 2024;8(2):144-8.
- [Background] Baghani P, Naserpour N, Piri H. Supervised Group Exercise Therapy Versus Home-based Exercise Therapy: The Effect of McGill Exercises on Pain, Disability and Trunk Stability in Middle-aged Women With Non-specific Chronic Low Back Pain. Physical Treatments-Specific Physical Therapy Journal. 2023;13(2):127-34.
- [Background] Aqil F, Iqbal MA, Karim S, Iqbal MU, Akram MJ, Mehreen Z, et al. Comparison of Mckenzie approach versus Lumbar Stabilization Exercises in the treatment of chronic low back pain. Rehman Journal of Health Sciences. 2021;3(1):24-31.
- [Background] Bose G, Gohill D. Effect of Mckenzie Therapy and Lumbar Strengthening Program in Lumbar Spine Derangement Syndrome 1. European Journal of Pharmaceutical and Medical Research. 2018;5(3):160-4.
- [Background] Namnaqani FI, Mashabi AS, Yaseen KM, Alshehri MA. The effectiveness of McKenzie method compared to manual therapy for treating chronic low back pain: a systematic review. Journal of musculoskeletal & neuronal interactions. 2019;19(4):492.
- [Background] Lam OT, Strenger DM, Chan-Fee M, Pham PT, Preuss RA, Robbins SM. Effectiveness of the McKenzie method of mechanical diagnosis and therapy for treating low back pain: literature review with meta-analysis. Journal of orthopaedic & sports physical therapy. 2018;48(6):476-90.
- [Background] Ghorbanpour A, Azghani MR, Taghipour M, Salahzadeh Z, Ghaderi F, Oskouei AE. Effects of McGill stabilization exercises and conventional physiotherapy on pain, functional disability and active back range of motion in patients with chronic non-specific low back pain. J Phys Ther Sci. 2018 Apr;30(4):481-485. doi: 10.1589/jpts.30.481. Epub 2018 Apr 13. PMID 29706690
- [Background] Olaoye MI, Okonji R, Ademoyegun A, Gebrye T, Yeowell G, Fatoye F, et al. Biochemical and clinical effects of McKenzie therapy versus muscle endurance exercises in chronic low-back pain. Arch Physiother. 2025;15:229-49.
- [Background] Calatayud J, Escriche-Escuder A, Cruz-Montecinos C, Andersen LL, Pérez-Alenda S, Aiguadé R, et al. Tolerability and muscle activity of core muscle exercises in chronic low-back pain. International journal of environmental research and public health. 2019;16(19):3509.
- [Background] Langevin HM, Sherman KJ. Pathophysiological model for chronic low back pain integrating connective tissue and nervous system mechanisms. Medical hypotheses. 2007;68(1):74-80.
- [Background] Casiano VE, Sarwan G, Dydyk AM, Varacallo MA. Back pain. StatPearls [Internet]: StatPearls Publishing; 2023.
- [Background] Mohd Isa IL, Teoh SL, Mohd Nor NH, Mokhtar SA. Discogenic low back pain: anatomy, pathophysiology and treatments of intervertebral disc degeneration. International journal of molecular sciences. 2022;24(1):208.
- [Background] Li W, Gong Y, Liu J, Guo Y, Tang H, Qin S, et al. Peripheral and central pathological mechanisms of chronic low back pain: a narrative review. Journal of pain research. 2021:1483-94.
- [Background] Borenstein D. Mechanical low back pain-a rheumatologist's view. Nature Reviews Rheumatology. 2013;9(11):643-53.
- [Background] Will JS, Bury DC, Miller JA. Mechanical Low Back Pain. Am Fam Physician. 2018 Oct 1;98(7):421-428. PMID 30252425
- [Background] Hnatešen D, Pavić R, Radoš I, Dimitrijević I, Budrovac D, Čebohin M, et al. Quality of Life and Mental Distress in Patients with Chronic Low Back Pain: A Cross-Sectional Study. International Journal of Environmental Research and Public Health. 2022;19(17):10657.
- [Background] Osagie RO, Tufa I, Angarita-Fonseca A, Pagé MG, Lacasse A, Stone LS, et al. Impact of different acute low back pain definitions on the predictors and on the risk of transition to chronic low back pain: a prospective longitudinal cohort study. PAIN. 2025;166(11):e577-e89.
- [Background] Nieminen LK, Pyysalo LM, Kankaanpää MJ. Prognostic factors for pain chronicity in low back pain: a systematic review. Pain reports. 2021;6(1):e919.